CLINICAL TRIAL: NCT02646800
Title: A Multi-center, Open-label, Non-comparative Study to Evaluate the Safety and Efficacy of Micafungin Against Fungal Infections Caused by Candida Spp or Aspergillus Spp
Brief Title: Post Marketing Study to Evaluate the Safety and Efficacy of Micafungin Against Fungal Infections Caused by Candida Spp or Aspergillus Spp
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to administrative reasons
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACN-MA-MYC-registry-2013
Record Dates: First submitted 2015-12-16; First posted 2016-01-06 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Aspergillosis; Candidiasis
Keywords: Micafungin; Antifungal; Candidiasis; Aspergillosis
MeSH Terms: conditions — Aspergillosis; Candidiasis | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Micafungin group (Experimental): Intravenous (IV)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — Injection

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of intravenous micafungin for the treatment of adult patients in China infected by Candida spp or Aspergillus spp.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed as proven/probable/possible fungal infection caused by Candida or Aspergillus based on the Chinese guidelines
* Females of childbearing potential must have a negative pregnancy test within 48 hrs prior to the study and reliable methods of contraception should be started 4 weeks prior to and during the whole study.
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study is obtained.
* Failure to fulfill inclusion criteria in another study, is not necessarily an exclusion criteria for this study, assuming other inclusion criteria 1-4 stated above are fulfilled.

Exclusion Criteria:

* Patient has history of hypersensitivity, or any serious reaction to any component of this product or other echinocandins.
* Subject is unlikely to comply with the visits scheduled in the protocol in the opinion of investigator or has a history of non-compliance.
* Pregnant women, nursing mothers, lactating women, and women of child-bearing potential who are unwilling to use reliable contraception for the duration of the study and for 6 weeks following completion of the study.
* AST/ALT > 5 times the upper limit of normal (ULN)
* Total bilirubin> 2.5 times ULN
* Patient has been previously enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03-21 (Actual); Primary Completion 2014-12-21 (Actual); Study Completion 2014-12-21 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by overall incidence and severity of adverse events for patients with candidiasis | Up to a maximum of 10 weeks
Safety as assessed by overall incidence and severity of adverse events for patients with aspergillosis | Up to a maximum of 14 weeks
Safety as assessed by adverse reactions for patients with candidiasis | Up to a maximum of 10 weeks
Safety as assessed by adverse reactions for patients with aspergillosis | Up to a maximum of 14 weeks

SECONDARY OUTCOMES:
Overall success rate for patients with candidiasis | End of treatment (up to up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis)
  Overall success rate=number of overall success patients/number of patients for efficacy evaluation × 100% at end of treatment (overall success is defined as patients with complete or partial response)
Overall success rate for patients with aspergillosis | End of treatment (up to 6 weeks, and up to 12 weeks for refractory patients)
  Overall success rate=number of overall success patients/number of patients for efficacy evaluation × 100% at end of treatment (overall success is defined as patients with complete or partial response)
Clinical Improvement rate for patients with candidiasis | End of treatment (up to up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis
Clinical Improvement rate for patients with aspergillosis | End of treatment (up to 6 weeks, and up to 12 weeks for refractory patients)
Fungal clearance rate for patients with candidiasis | End of treatment (up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis)
Fungal clearance rate for patients with aspergillosis | End of treatment (up to 6 weeks, and up to 12 weeks for refractory patients
Fatality rate for patients with candidiasis | End of treatment (up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis)
Fatality rate for patients with aspergillosis | End of treatment (up to 6 weeks, and up to 12 weeks for refractory patients
Safety as assessed by relationship of adverse events to Micafungin for patients with candidiasis | Day 1 to the end of treatment (up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis)
Safety as assessed by relationship of adverse events to Micafungin for patients with aspergillosis | Day 1 to the end of treatment (up to 6 weeks, and up to 12 weeks for refractory patients)
Safety as assessed by liver and kidney function for patients with candidiasis | Day 1 to the end of treatment (up to 4 weeks, and up to 8 weeks for patients with chronic disseminated candidiasis, candida osteomyelitis, or candida endocarditis)
Safety as assessed by liver and kidney function for patients with aspergillosis | Day 1 to the end of treatment (up to 6 weeks, and up to 8 weeks, and up to 12 weeks for refractory patients)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (16):
- China (16):
  - Beijing
  - Changchun
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Harbin
  - Hengyang
  - Jinan
  - Nanjing
  - Qingdao
  - Shijiazhuang
  - Taiyuan
  - Tianjing
  - Ürümqi
  - Xi'an

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results Web site — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=ACN-MA-MYC-registry-2013